CLINICAL TRIAL: NCT06216808
Title: A Prospective, Multicenter, Single Arm, Open Label, First-in-human Study to Evaluate the Safety and Initial Efficacy of HyperQureTM, Laparoscopic Renal Denervation Therapy, in Patients With Resistant Hypertension on 3 or More Antihypertensive Medications
Brief Title: A First-in-human Study of HyperQureTM", Laparoscopic Renal Denervation Therapy in Patient With Resistant Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DeepQure Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HQ-HTN-K01-02
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Intervention Model Description: The HyperQure RDN System consists of a generator that generates RF(Radiofrequency) energy and a Laparoscopic Instrument that delivers the RF energy generated by the generator to the treatment area. Through a laparoscopic approach, the renal artery is accessed through the retroperitoneum, which is the closest path to the renal artery. After wrapping 360 degrees of renal artery, RDN is performed as per the preset parameters of 50 degrees and 70 seconds. The target blood vessel is planned by CTA before the procedure, and the proximal and distal areas of the right and left main renal artery are treated once at a distance of at least 3 mm respectively, and RDN is also performed on the branch or accessory vessel confirmed to be suitable for the procedure by CTA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Laparoscopic Renal Denervation (Experimental): Intervention:
  Device: HyperQure Renal Denervation System
  Interventions: Device: HyperQure Renal Denervation System

INTERVENTIONS:
Device: HyperQure Renal Denervation System — The HyperQure RDN System consists of a generator that generates RF energy and a Laparoscopic Instrument that delivers the RF energy generated by the generator to the treatment area. Through a laparoscopic approach, the renal artery is accessed through the retroperitoneum, which is the closest path to the renal artery. After wrapping 360 degrees of renal artery, RDN is performed as per the preset parameters of 50 degrees and 70 seconds.
  The target blood vessel is planned by CTA before the procedure, and the proximal and distal areas of the right and left main renal artery are treated once at a distance of at least 3 mm respectively, and RDN is also performed on the branch or accessory vessel confirmed to be suitable for the procedure by CTA.

SUMMARY:
HQ-HTN-K01-02 is a prospective, multicenter, single arm, open label, first-in-human study to evaluate the safety and initial efficacy of HyperQureTM, laparoscopic denervation therapy, in patients with resistant hypertension on 3 or more antihypertensive medications

DETAILED DESCRIPTION:
< Study purpose > The purpose of this single arm interventional study is to evaluate the safety and initial efficacy of HyperQureTM, laparoscopic renal denervation therapy, in patients with resistant hypertension on 3 or more antihypertensive medications including a diuretic

< Background and Hypothesis > The HyperQureTM RDN(Renal Denervation) System is developed to overcome the limitations of endovascular RDN using catheters; 1)incomplete renal denervation, 2) risk of intimal damage due to intravascular access, and 3) access limitations due to vascular anatomy and size The HyperQureTM RDN System is accessed through the adventitia where renal sympathetic nerves are mainly distributed. Since energy is transmitted by wrapping the blood vessel 360 degrees, it is expected that it will be possible to achieve more complete renal denervation, reduce the risk of intimal damage, and solve structural access problems caused by the anatomy and size of the renal blood vessel.

< Study plan > Ten eligible adult men and women with resistant hypertension will be enrolled and will have laparoscopic RDN under general anesthesia.

CTA(Computed Tomographic Angiogram), blood tests, office blood pressure, 24-hour ambulatory blood pressure and QOL will be monitored to evaluate the safety and initial efficacy for 12 months after RDN procedure.

ELIGIBILITY:
Inclusion Criteria:

Subjects are deemed eligible for this clinical trial only if they meet all of the following criteria:

1. Male and female patients aged between 19 and 79 years old
2. Resistant hypertensive patients on stable regimen of at least 3 antihypertensive medications* for at least 4weeks prior Screening1 and those who are willing to continue existing antihypertensive medications during run- in period and till 3 months after surgery from Screening 1

   * Patients on at least 3 antihypertensive medications of different classes including diuretics
3. Those who meet the following blood pressure requirements:

   [Screening 1]
   * Office systolic blood pressure (SBP) ≥ 140 mmHg
   * Office diastolic blood pressure (SBP) ≥ 90 mmHg

   [Screening 2]
   * Office SBP ≥ 140 mmHg
   * Office DBP ≥ 90 mmHg
   * Daytime ASBP ≥ 135 mmHg
4. Those who have the ability and willingness to provide voluntary and written consent to participate in this clinical trial

Exclusion Criteria:

Subjects cannot be enrolled in the clinical trial if they meet any of the following criteria

1. Those with the following confirmed anatomical findings in the kidney or renal artery that are unsuitable for renal denervation (assessed based on the results of the renal CT angiography of Screening 2)

   * If there is an atheroma or renal artery stent within 5 mm of the renal denervation site
   * Presence of stenosis of 30% or more on all of the blood vessels available for renal denervation therapy
   * When it is deemed impossible to perform denervation on both renal arteries according to the discretion of the investigator
2. Those with a medical history or a history of surgery/procedure that is unsuitable for renal denervation therapy

   * Renal denervation therapy
   * Renal artery stenting within 3 months prior to surgery
   * Polycystic kidney disease (PKD)
   * Atrophic kidney
   * Kidney transplant
   * Dialysis due to end-stage renal disease
   * Any surgery performed on the both kidney
   * FMD(Fibromuscular dysplasia)
3. Those with a confirmed comorbidity or a history of surgery/procedure that is unsuitable for posterior retroperitoneal approach required for renal denervation therapy

   * Surgical history using the retroperitoneal approach
   * Fibrosis of the retroperitoneal region
   * Inflammation of the retroperitoneal region
   * Extreme obesity (body mass index (BMI) > 40 kg/m2)
   * Risk of elevated intracranial pressure
4. eGFR* < 45 mL/min/1.73 m2

   * eGFR calculation formula (MDRD equation) 175 × (sCr)-1.154 × (age)-0.203 × (0.742 if female)
5. Those with type 1 diabetes or uncontrolled type 2 diabetes*

   * Uncontrolled type 2 diabetes: HbA1c ≥ 8.0%
   * HbA1c will be tested in Screening 2 if the confirmed HbA1c result is from the test conducted 3 months before Screening 2 or if additional tests are deemed necessary according to the investigator discretion due to a history of inadequately controlled blood glucose level.
6. Those who receive SGLT2 inhibitors or GLP-1 agonists within 90 days before Screening 1, or those who are expected to require treatment during the clinical trial period(but if on continuous medication without changes more than 90days can be enrolled)
7. Those with at least a 20-mmHg decrease in office SBP or at least a 10-mmHg decrease in office DBP accompanied by symptoms, measured within 3 minutes of standing up during Screening 2(but if orthostatic hypotension is clearly due to Benign Prostatic Hyperplasia, subject can be enrolled)
8. Those who are likely to experience safety problems due to blood pressure drop according to the discretion of the investigator (e.g., heart valve stenosis, peripheral vascular disease, aortic aneurysm, and high-risk groups for bleeding (thrombocytopenia, hemophilia, severe anemia, etc.)
9. Those who have difficulty in measuring blood pressure accurately according to the discretion of the investigator (e.g., if the circumference of the upper arm is larger than the cuff size of the blood pressure monitor, those with arrhythmia, etc.)
10. Those who have secondary hypertension or are receiving sympathomimetic drugs that affect hypertension
11. Those with a history of the following cardiovascular diseases or accompanying diseases

    * Myocardial infarction occurring within 3 months prior to Screening 1
    * Stable/Unstable angina occurring within 3 months prior to Screening 1
    * Heart failure(NYHA classification III~IV) within 3 months prior to Screening 1
    * Transient ischemic attack within 3 months prior to Screening 1
    * Cerebrovascular seizures (e.g., subarachnoid hemorrhage, cerebral embolism, etc.) within 3 months prior to Screening 1
    * Atrial fibrillation (except for those who have confirmed sinus rhythm after undergoing medicinal treatment or surgery such as catheterization for the treatment of atrial fibrillation)
12. Those with primary pulmonary hypertension
13. Those with confirmed bleeding diathesis, coagulation disorder, or refusal to receive transfusions
14. Those with a history of peptic ulcer disease or gastrointestinal bleeding within 6 months prior to Screening 1
15. Those who are chronically on oxygen-assisted or mechanical ventilation (e.g., CPAP, BiPAP) (however, usage due to sleep apnea is exempted)
16. Those who have taken non-steroidal anti-inflammatory drugs (NSAIDs) twice or more per week for pain control within 1 month prior to Screening 2
17. Those with a history of contraindications to the use of contrast agents, anaphylactic reactions, or uncontrolled allergic reactions
18. Those receiving antiretroviral drug therapy due to HIV infection (except when there is a documented history of hypertension prior to initiation of antiretroviral drug therapy)
19. Those with the following confirmed drug administration history in relation to narcotic drugs:

    * A history of abuse of narcotic drugs
    * Those who use methadone
    * Those who have used narcotic drugs twice or more within 1 month prior to Screening 1
20. Those with drug or alcohol dependence that has not been cured at the time of Screening 1, and who lack the ability or are unable to understand and follow the instructions required in this clinical trial
21. Those who are scheduled to undergo a surgery/procedure that is expected to affect the efficacy and safety of this clinical trial according to the discretion of the investigator
22. Night shift workers
23. Those who have received other investigational products or investigational medical devices within 4 weeks prior to Screening 1 (however, such patients may be enrolled if such products of devises do not affect the efficacy and safety assessment of this clinical trial according to the discretion of the investigator)
24. Women who are pregnant, lactating, or plan to become pregnant during the period of the clinical trial
25. Other subjects who are deemed ineligible to participate in this clinical trial according to the investigator's discretion

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Change in 24-h Ambulatory Systolic Blood Pressure(ASBP) | from baseline to 3 months post procedure
  Change in 24-h ASBP from baseline at 3 months post procedure

SECONDARY OUTCOMES:
Change in 24-h ASBP | from baseline to 6, 12 months post procedure
  Change in 24-h ASBP from baseline to 6, 12 months post procedure
Change in 24-h Ambulatory Diastolic Blood Pressure(ADBP) | from baseline to 3, 6, 12 months post procedure
  Change in 24-h ADBP from baseline to 3, 6, 12 months post procedure
Change in daytime ASBP and ADBP | from baseline to 3, 6, 12 months post procedure
  Change in daytime ASBP and ADBP from baseline to 3, 6, 12 months post procedure
Change in nighttime ASBP and ADBP | from baseline to 3, 6, 12 months post procedure
  Change in nighttime ASBP and ADBP from baseline to 3, 6, 12 months post procedure
Change in Office Systolic Blood Pressure(SBP) and Diastolic Blood Pressure(DBP) | from baseline to 1, 3, 6, 12 months post-procedure
  Change in office SBP and DBP from baseline to 1, 3, 6, 12 months post procedure
Incidence of achieving target office SBP (SBP <140 mmHg) | at 1, 3, 6, 12 months post-procedure
  Incidence of achieving target office SBP(SBP <140mmHg) at 1, 3, 6, 12 months post procedure
Change in EQ-5D from baseline | at 3, 6, 12 months post procedure
  Change in EQ-5D from baseline at 3, 6, 12 months post procedure. EQ-5D-5L is a QOL(Quality of Life) evaluation tool. This includes a "Questionnaire of five dimensions" to evaluate mobility, self-care, usual activities, discomfort or pain and depression or anxiety scored from level 1 to 5 (lower level means a better outcome; ex. level 1 of Mobility is "I have no problems in walking about) and also includes "EQ VAS" to evaluate "YOUR HEALTH TODAY" and this scale is numbered from 0 to 100.
Incidence and patterns of adverse events | from baseline to 3 and 12 months post procedure
  Incidence and patterns of adverse events from baseline to 3 and 12 months post procedure
Incidence of major adverse events (MAE)* | from baseline to 1, 3, 6 and 12 months post procedure
  * MAE
  * All deaths
  * End-stage renal disease
  * Severe embolism resulting in end-organ damage
  * Renal artery dissection requiring intervention
  * Renal artery perforation requiring intervention
  * Vascular complications
  * Hypertensive crisis requiring hospitalization (unless due to non-compliance with drugs or therapy)
  * Newly confirmed renal artery stenosis (>70%)
Incidence of each of the following acute/procedural adverse event | from baseline to 1 month post procedure
  * Postoperative complications rated as grade 3 or higher according to the Clavien-Dindo classification
  * Severe embolism resulting in end-organ damage
  * Renal artery dissection requiring intervention
  * Renal artery perforation requiring intervention
  * Vascular complications
  * End-stage renal disease
  * Hypertensive crisis requiring hospitalization (unless due to non-compliance with drugs or therapy)
  * Decrease in eGFR (≥40%)
  * Newly confirmed myocardial infarction
  * Newly confirmed stroke
  * Renal artery reoperation/surgery
  * Major bleeding in thrombolysis in myocardial infarction (TIMI)*
    * Death due to intracranial hemorrhage, absolute decrease in hemoglobin ≥5 g/m or in hematocrit ≥15%, or bleeding occurring within 7 days of surgery
  * More than 50% reduction in serum creatinine compared to Screening 2
  * Newly confirmed renal artery stenosis (>70%)
Incidence of each of the following adverse events | from baseline to 3, 6 and 12 months post procedure
  * All deaths
  * Newly confirmed renal artery stenosis (>70%)
  * End-stage renal disease
  * Hypertensive crisis requiring hospitalization (unless due to non-compliance with drugs or therapy)
  * Decrease in eGFR (≥40%)
  * Newly confirmed myocardial infarction
  * Newly confirmed stroke
  * Renal artery reoperation/surgery
  * Major bleeding in thrombolysis in myocardial infarction (TIMI)*
    * Death due to intracranial hemorrhage, absolute decrease in hemoglobin ≥5 g/mL or in hematocrit ≥15%, and bleeding occurring within 7 days of surgery
  * More than 50% reduction in serum creatinine compared to Screening 2
Normal/Abnormal conversion rate of laboratory test results | from baseline to 1, 3, 6 and 12 months post procedure
  Normal/Abnormal conversion rate of laboratory test results from baseline to 1, 3, 6 and 12 months post procedure
Change in heart rate | from baseline to 1, 3, 6 and 12 months post procedure
  Change in heart rate from baseline to 1, 3, 6 and 12 months post procedure

OTHER OUTCOMES:
Change in antihypertensive medication usage throughout the study | from baseline to 12 months post procedure
  Change in antihypertensive medication usage from baseline to 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: SungHoo Hong, MD, Principal Investigator — The Catholic University of Korea
Locations (7):
- South Korea (7):
  - Chonnam National University Hospital Hwasun Hospital, Jeonam, Chonnam Province
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No